CLINICAL TRIAL: NCT04911387
Title: iCare® Home vs Goldmann Applanation Tonometry: Agreement of the Methods and Comparison of Inter-observer Variation at a Tertiary Eye Centre
Brief Title: iCare® Home vs Goldmann Applanation Tonometry
Status: Completed | Type: Observational
Sponsor: St. Erik Eye Hospital (Other)
Responsible Party: Principal Investigator, Enping Chen, MD Ph D, St. Erik Eye Hospital
Other Study IDs: iCare Home vs GAT
Record Dates: First submitted 2021-05-18; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Glaucoma; Open Angle Glaucoma; Ocular Hypertension; Pseudo Exfoliation Syndrome
Keywords: intraocular pressure; GAT; rebound tonometry; self-tonometry; iCare® Home
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Ocular Hypertension; Exfoliation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Intraocular pressure measurments — Intraocular pressure measurements with iCare Home by participants (patients, volunteers) and healthcare staff as well as intraocular pressure measurements with GAT by participants different healthcare staff.

SUMMARY:
Self-tonometry with iCare Home is regularly performed at Sankt Erik's Eye Hospital since a few years back. The purpose of this study was to show that the eye pressure measurements made with iCare® Home by patients / relatives do not vary more than those made with the standard method, Goldman applanation tonometry (GAT), by different healthcare professionals. This will hopefully confirm the usefulness of self-tonometry.

DETAILED DESCRIPTION:
Since a few years back, self-tonometry with iCare® Home has been available in glaucoma care. Sankt Erik's Eye Hospital was first in Sweden to use the new technology. Several studies have shown good agreement between measurements made by patients or healthcare professionals with iCare® Home and Goldman applanation tonometry (GAT). However, some researchers raise critical voices about the reliability of iCare® Home measurements because they can differ from GAT. GAT is considered the gold standard method of tonometry to which all other instruments are compared. But like all other methods, GAT has some limitations.

At the clinic, the eye pressure is usually measured with GAT by different staff (ophthalmological nurses, opticians or doctors) from visit to visit. This can sometimes lead to pressure variations that may affect the follow-up of glaucoma patients. This raises the question of whether the difference between GAT and iCare® Home is statistically and clinically significant.

The purpose of this study was to show that the eye pressure measurements made with iCare® Home by patients / relatives do not vary more than those made with the standard method GAT by different healthcare professionals. This will hopefully confirm the usefulness of self-tonometry.

ELIGIBILITY:
Inclusion Criteria:

* primary open angle glaucoma (POAG)
* pseudo-exfoliation glaucoma (PEX)
* ocular hypertension (OHT)
* no eye disease,

Exclusion Criteria:

* inability to perform measurements due to limited hand or arm mobility (eg rheumatism, tremor)
* measurements outside the iCare® Home manufacturer's recommendations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who are referred to the clinic to perform a Eye pressure curve with iCare® Home are offered to participate in the study. The patient him-/herself or someone accompanying him/her may perform the measurements. Volunteer without an eye history to participate.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Correlation between iCare® Home inter-user measurements | 12 months
  iCare® Home measurements made by participants (patients and volunteers) will be compared to iCare® Home measurements made by trainers' using the same device on the same occasion
Correlation between GAT measurements made by different healthcare personnel | 12 months
  GAT measurements made by iCare® Home trainers will be compared to GAT measurements made by other available healthcare personnel using a different device on the same occasion

SECONDARY OUTCOMES:
Agreement between iCare® Home tonometry and GAT | 12 months
  Agreement, repeatability and reliability of measurements made with iCare® Home tonometry and GAT will be assessed using Bland Altman analysis, ANOVA and interclass correlation coefficient (ICC).

CONTACTS AND LOCATIONS:
Overall Officials: Enping Chen, MD Ph D, Principal Investigator — St. Erik Eye Hospital
Locations (1):
- St Erik Eye Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No